CLINICAL TRIAL: NCT06813950
Title: IMPACT of a PHYSICAL ACTIVITY PROGRAM on the HEALTH-RELATED QUALITY of LIFE in PEDIATRIC CANCER PATIENTS
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sociedad de Lucha Contra el Cáncer (Other)
Responsible Party: Principal Investigator, Gustavo Galarraga, Analyst Investigation Department, Sociedad de Lucha Contra el Cáncer del Ecuador
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2024-068M
Record Dates: First submitted 2025-02-03; First posted 2025-02-07 (Actual); Last update posted 2025-02-11 (Actual); Status verified 2025-02

CONDITIONS: Cancer; Pediatric Cancer
Keywords: physical activity; Quality of life; physical activity programs; lifestyle
MeSH Terms: conditions — Neoplasms; Motor Activity | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Physical activity (Other): Performs supervised physical activity
  Interventions: Other: Physical activity

INTERVENTIONS:
Other: Physical activity — The intervention group will participate in a 10-week structured physical activity program consisting of 120 minutes of supervised exercise per week, led by a team of physiotherapists and physical activity professionals. Meanwhile, the control group will not participate in any organized physical activity program but will continue with their usual activities.

SUMMARY:
Physical activity is essential for the health and well-being of children and adolescents. However, those living with cancer often experience reduced physical activity levels, which negatively impact their functional capacity and health-related quality of life (HRQoL). In Ecuador, data from the National Institute of Statistics and Census (2021) reveal that 20% of children engage in less than one hour of physical activity per week, highlighting the need for targeted interventions. While previous studies demonstrate that supervised exercise programs can improve physical and psychosocial health outcomes in pediatric oncology patients, no evidence exists from Ecuador to assess the effects of such programs.

This study will examine the impact of a structured physical activity program on the HRQoLof pediatric cancer patients in Quito, Ecuador. Using a case-control design, 90 participants will be randomized into two groups: an intervention group receiving a 10-week, supervised physical activity program and a control group with no exercise intervention and the programmed usual care as follow up if needed by the social worker. HRQoL surveys using a standardized instrument will be administered to all participants (those in the intervention group and those in the control group) at weeks 1, 12, and 24 to assess changes over time.

This research will address a critical public health gap by exploring how physical activity can mitigate the adverse effects of cancer treatment, improve physical and emotional health, and enhance the HRQoL in pediatric oncology patients. Findings will contribute valuable insights for integrating physical activity into pediatric oncology care in low- and middle-income countries.

DETAILED DESCRIPTION:
This study is designed as a randomized controlled trial (RCT) to investigate the impact of a structured exercise program on the HRQoL of pediatric cancer patients. A total of 90 participants will be recruited and randomly assigned to either the intervention group or the control group.

The intervention group will participate in a 10-week structured physical activity program consisting of 120 minutes of supervised exercise per week, led by a team of physiotherapists and physical activity professionals. Meanwhile, the control group will not participate in any organized physical activity program but will continue with their usual activities.

Both groups will complete the Pediatric Quality of Life Inventory (PedsQL) surveys at baseline (week 1), midpoint (week 12), and endpoint (week 24). These surveys are designed to assess changes in participants' HRQoL over time, providing comparative insights between the two groups.

ELIGIBILITY:
Inclusion Criteria:

* 1. Age range: Participants must be between 8 and 18 years old at the start of the study.

  2. Residency: Patients residing within the city limits of Quito, Ecuador. 3. Treatment status:

  • Patients are being evaluated or treated at Hospitals SOLCA and Baca Ortiz.
  * Patients are either currently undergoing active treatment for pediatric malignancies, or
  * Patients are in the post-treatment phase after a pediatric cancer diagnosis.
  * The volunteer or a family member that lives with the possible participant has a cellphone so the survey can be administered and answered.

Exclusion Criteria:

* 1. The presence of a malignant solid tumor which has not yet been surgically addressed.

  2. A psychiatric diagnosis of cognitive impairment. 3. A diagnosis of osteosarcoma. 4. A history of cardiac pathology. 5. The patient is in the pediatric inpatient ward or was one month prior to the enrollment phase.

  6. The patient is stationed at the pediatric intensive care unit. 7. The patient received high-dose chemotherapy with methotrexate greater than 1000 mg/m2/dose or cytarabine greater than 1 g/m2/dose in the last month.

Ages: 8 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 80 (Estimated)
Dates: Start 2025-02-20 (Estimated); Primary Completion 2025-11 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Health related quality of life | oth groups will complete the Pediatric Quality of Life Inventory (PedsQL) surveys at baseline (week 1), midpoint (week 12), and endpoint (week 24). These surveys are designed to assess changes in participants' HRQoL over time, providing comparative insig
  To evaluate HRQoL, the study will use the PedsQL, specifically the PedsQL 3.0 Cancer Module, a validated instrument for pediatric cancer patients aged 2 to 18 years. This module comprises 20 questions addressing physical, emotional, and social functioning, as well as cancer treatment-related symptoms. Participants will self-report their responses using a four-point Likert scale, with options ranging from "never" (0) to "almost always" (4). For example: "In the past month, how often have you felt tired?"; "In the past month, how often have you experienced pain or discomfort?".

SECONDARY OUTCOMES:
Physical activity | surveys at baseline (week 1), midpoint (week 12), and endpoint (week 24).
  Physical activity and sedentary habits will be determined using the Activity Profile - Spain - Version for Latin America. (YAP-SL), a self-report tool consisting of 15 items, will be used to gather data on physical activity levels and sedentary behaviors for a 7-day recall period

CONTACTS AND LOCATIONS:
Overall Officials: Gustavo Galárraga, MPH, Principal Investigator — Sociedad de Lucha Contra el Cáncer
Locations (1):
- SociedadLuchaContraCáncer, Quito, Pichincha, Ecuador

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Varni JW, Burwinkle TM, Katz ER, Meeske K, Dickinson P. The PedsQL in pediatric cancer: reliability and validity of the Pediatric Quality of Life Inventory Generic Core Scales, Multidimensional Fatigue Scale, and Cancer Module. Cancer. 2002 Apr 1;94(7):2090-106. doi: 10.1002/cncr.10428. PMID 11932914
- [Background] Segura-Diaz JM, Barranco-Ruiz Y, Saucedo-Araujo RG, Aranda-Balboa MJ, Cadenas-Sanchez C, Migueles JH, Saint-Maurice PF, Ortega FB, Welk GJ, Herrador-Colmenero M, Chillon P, Villa-Gonzalez E. Feasibility and reliability of the Spanish version of the Youth Activity Profile questionnaire (YAP-Spain) in children and adolescents. J Sports Sci. 2021 Apr;39(7):801-807. doi: 10.1080/02640414.2020.1847488. Epub 2020 Nov 20. PMID 33213295
- [Background] Saint-Maurice PF, Welk GJ. Validity and Calibration of the Youth Activity Profile. PLoS One. 2015 Dec 2;10(12):e0143949. doi: 10.1371/journal.pone.0143949. eCollection 2015. PMID 26630346
- [Background] de Onis M, Onyango AW, Borghi E, Siyam A, Nishida C, Siekmann J. Development of a WHO growth reference for school-aged children and adolescents. Bull World Health Organ. 2007 Sep;85(9):660-7. doi: 10.2471/blt.07.043497. PMID 18026621
- [Background] Riedl D, Licht T, Nickels A, Rothmund M, Rumpold G, Holzner B, Grote V, Fischer MJ, Fischmeister G. Large Improvements in Health-Related Quality of Life and Physical Fitness during Multidisciplinary Inpatient Rehabilitation for Pediatric Cancer Survivors. Cancers (Basel). 2022 Oct 4;14(19):4855. doi: 10.3390/cancers14194855. PMID 36230777
- [Background] Keats MR, Culos-Reed SN. A community-based physical activity program for adolescents with cancer (project TREK): program feasibility and preliminary findings. J Pediatr Hematol Oncol. 2008 Apr;30(4):272-80. doi: 10.1097/MPH.0b013e318162c476. PMID 18391695
- [Background] Gotte M, Taraks S, Boos J. Sports in pediatric oncology: the role(s) of physical activity for children with cancer. J Pediatr Hematol Oncol. 2014 Mar;36(2):85-90. doi: 10.1097/MPH.0000000000000101. PMID 24390449
- [Background] Rapti C, Dinas PC, Chryssanthopoulos C, Mila A, Philippou A. Effects of Exercise and Physical Activity Levels on Childhood Cancer: An Umbrella Review. Healthcare (Basel). 2023 Mar 10;11(6):820. doi: 10.3390/healthcare11060820. PMID 36981477
- [Background] Chaput JP, Willumsen J, Bull F, Chou R, Ekelund U, Firth J, Jago R, Ortega FB, Katzmarzyk PT. 2020 WHO guidelines on physical activity and sedentary behaviour for children and adolescents aged 5-17 years: summary of the evidence. Int J Behav Nutr Phys Act. 2020 Nov 26;17(1):141. doi: 10.1186/s12966-020-01037-z. PMID 33239009
- [Background] Zhang FF, Saltzman E, Must A, Parsons SK. Do Childhood Cancer Survivors Meet the Diet and Physical Activity Guidelines? A Review of Guidelines and Literature. Int J Child Health Nutr. 2012;1(1):44-58. doi: 10.6000/1929-4247.2012.01.01.06. Epub 2012 Sep 25. PMID 26973721
- [Background] Braam KI, van der Torre P, Takken T, Veening MA, van Dulmen-den Broeder E, Kaspers GJ. Physical exercise training interventions for children and young adults during and after treatment for childhood cancer. Cochrane Database Syst Rev. 2013 Apr 30;(4):CD008796. doi: 10.1002/14651858.CD008796.pub2. PMID 23633361
- [Background] Oficina Regional para las Américas de la Organización Mundial de la Salud. https://www.paho.org/es/temas/cancer-ninez-adolescencia#:~:text=En%20Am%C3%A9rica%20Latina%20y%20el,a%20causa%20de%20esta%20enfermedad. 2014 [cited 2024 Dec 1]. EL CÁNCER INFANTIL EN LAS AMÉRICAS. Available from: https://www.paho.org/es/temas/cancer-ninez-adolescencia#:~:text=En%20Am%C3%A9rica%20Latina%20y%20el,a%20causa%20de%20esta%20enfermedad
- [Background] San Juan AF, Chamorro-Vina C, Mate-Munoz JL, Fernandez del Valle M, Cardona C, Hernandez M, Madero L, Perez M, Ramirez M, Lucia A. Functional capacity of children with leukemia. Int J Sports Med. 2008 Feb;29(2):163-7. doi: 10.1055/s-2007-964908. Epub 2007 Sep 18. PMID 17879894
- [Background] Tillmann V, Darlington AS, Eiser C, Bishop NJ, Davies HA. Male sex and low physical activity are associated with reduced spine bone mineral density in survivors of childhood acute lymphoblastic leukemia. J Bone Miner Res. 2002 Jun;17(6):1073-80. doi: 10.1359/jbmr.2002.17.6.1073. PMID 12054163
- [Background] 3. INEC. Juntos para combatir el sedentarismo mediante el deporte y la actividad física. 2022. Juntos para combatir el sedentarismo mediante el deporte y la actividad física.
- [Background] Wurz A, McLaughlin E, Lategan C, Chamorro Vina C, Grimshaw SL, Hamari L, Gotte M, Kesting S, Rossi F, van der Torre P, Guilcher GMT, McIntyre K, Culos-Reed SN. The international Pediatric Oncology Exercise Guidelines (iPOEG). Transl Behav Med. 2021 Oct 23;11(10):1915-1922. doi: 10.1093/tbm/ibab028. PMID 34037786